CLINICAL TRIAL: NCT04071613
Title: Tenecteplase Versus Alteplase for Stroke Thrombolysis Evaluation Trial in the Ambulance
Acronym: TASTEa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.043
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-10

CONDITIONS: Stroke, Acute, Stroke Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomised open-label blinded endpoint (PROBE) phase II study in stroke thrombolysis patients to compare tenecteplase and alteplase for an outcome of less disability at 3 months
Who Masked: Outcomes Assessor
Masking Description: The people assessing the outcomes The people analysing the results/data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous tenecteplase (TNK) (Active Comparator): Patients will receive intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over ~10 seconds).
  Interventions: Drug: Tenecteplase
- Intravenous tissue plasminogen activator (tPA) (Active Comparator): Patients will receive intravenous t-PA at the standard licensed dose of 0.9 mg/kg up to a maximum of 90mg, 10% as bolus and the remainder over 1 hour.
  Interventions: Drug: Intravenous tissue plasminogen activator (tPA)

INTERVENTIONS:
Drug: Tenecteplase — Route: IV bolus injection Frequency: once only, within 4.5 hours of stroke onset
  Other Names: TNK
  Arms: Intravenous tenecteplase (TNK)
Drug: Intravenous tissue plasminogen activator (tPA) — Route: Intravenous (IV) infusion (10% as bolus and the remainder over 60 minutes) Frequency: once only, within 4.5 hours of stroke onset
  Other Names: TPA, Alteplase
  Arms: Intravenous tissue plasminogen activator (tPA)

SUMMARY:
Ischemic stroke is a major health burden globally and in Australia. Treatment for ischemic stroke is time critical and is significantly more effective if administered within the first 90 minutes of symptom onset. This clinical trial will identify if early administration of oral thrombolytic agent, tenecteplase prior to hospital can improve outcomes from stroke, and reduce costs compared to standard care of IV alteplase in hospital

DETAILED DESCRIPTION:
Currently, alteplase is the standard clot-dissolving therapy for ischemic stroke, however this treatment is only effective in 30-45% of patients. Importantly, treatment of ischemic stroke is more effective when given within 90 minutes of stroke onset. Means of treating patients earlier with more effective therapies are needed.

Ischemic stroke is a major public health problem, for which effective and accessible drug therapies remain limited. Current management of acute ischemic stroke includes treatment with a solution called alteplase, which dissolves clots in a cerebral artery. The treatment effect of alteplase is much greater if given within 90 minutes of stroke onset.

As a result, there has been a significant push to take stroke care to the patient in the form of the Mobile Stroke Unit (MSU). The MSU is the first designed as a CT-capable ambulance that allows assessment and treatment of stroke patients in the pre-hospital setting. In the proposed research project, we will undertake a clinical trail investigating the effectiveness of a new thrombolytic agent in the MSU, tenecteplase.

Tenecteplase has been shown to be significantly more effective at improving stroke survivor's recovery and opening blocked blood vessels than alteplase in the hospital setting. However, it is unknown if earlier administration of tenecteplase is more effective than early administration of alteplase.

The tested agent, tenecteplase, is cheaper, easier to administer (no time-consuming infusions required) and more practical for an ambulance delivered therapy than the current standard of care alteplase. If tenecteplase results in better clinical outcomes in addition to these practical advantages, there is significant scope for improved patient outcomes and cost savings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients being attended by the mobile stroke unit with an acute ischemic stroke eligible for thrombolysis using standard clinical and CT criteria.
2. Patient's age is ≥18 years
3. Premorbid mRS <4

Exclusion Criteria:

1. Intracranial hemorrhage (ICH) or other diagnosis (e.g. tumor) identified by CT on the MSU
2. Hypodensity in >1/3 MCA territory or equivalent proportion of ACA or PCA territory on non-contrast CT on MSU
3. Pre-stroke mRS score of > 3 (indicating significant previous disability)
4. Any terminal illness such that patient would not be expected to survive more than 1 year
5. Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
6. Pregnant women.
7. Rapidly improving symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Perfusion lesion on CTP | Within 2hrs of treatment
  The volume of the perfusion lesion on CTP performed on arrival at the receiving hospital, adjusted for pre-treatment NIHSS and time from initiation of treatment to CTP.

SECONDARY OUTCOMES:
Infarct core growth between baseline CTP and 24 hour MRI. | 24 hrs
Percent reperfusion between baseline CTP and 24 hour perfusion imaging (MRI) | 24 hrs
Reduction in NIHSS between pre-treatment score and score on ED arrival, adjusted for pre-treatment NIHSS and time from initiation of treatment to ED NIHSS score | 2 hrs
Reduction in NIHSS between pre-treatment score and score at 24 hours post treatment, adjusted for pre-treatment NIHSS | 24 hrs
Modified Rankin Scale (mRS) at 3 months - ordinal analysis adjusted for baseline NIHSS and age | 3 months
mRS 0-2 or no change from baseline at 3 months adjusted for baseline NIHSS and age | 3 months
Proportion of patients where thrombolytic medication is initiated within 5 minutes of completion of CT on the MSU. | 24 hrs
Time from completion of CT on the MSU to initiation of thrombolysis (CT to needle time) | 2 hrs
mRS 5-6 at 3 months adjusted for baseline NIHSS and age | 3 months
Death due to any cause adjusted for baseline NIHSS and age | During time on study up to 3 months
Any parenchymal haematoma | During time on study up to 3 months
ymptomatic intracranial hemorrhage (sICH) | During time on study up to 3 months

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Eastern Health, Melbourne, Victoria
  - Western Hospital, Melbourne, Victoria
  - Alfred Hopsital, Melbourne
  - Monash Health, Melbourne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bivard A, Zhao H, Churilov L, Campbell BCV, Coote S, Yassi N, Yan B, Valente M, Sharobeam A, Balabanski AH, Dos Santos A, Ng JL, Yogendrakumar V, Ng F, Langenberg F, Easton D, Warwick A, Mackey E, MacDonald A, Sharma G, Stephenson M, Smith K, Anderson D, Choi P, Thijs V, Ma H, Cloud GC, Wijeratne T, Olenko L, Italiano D, Davis SM, Donnan GA, Parsons MW; TASTE-A collaborators. Comparison of tenecteplase with alteplase for the early treatment of ischaemic stroke in the Melbourne Mobile Stroke Unit (TASTE-A): a phase 2, randomised, open-label trial. Lancet Neurol. 2022 Jun;21(6):520-527. doi: 10.1016/S1474-4422(22)00171-5. Epub 2022 May 4. PMID 35525251
- [Derived] Bivard A, Zhao H, Coote S, Campbell B, Churilov L, Yassi N, Yan B, Valente M, Sharobeam A, Balabanski A, Dos Santos A, Ng F, Langenberg F, Stephenson M, Smith K, Bernard S, Thijs V, Cloud G, Choi P, Ma H, Wijeratne T, Chen C, Olenko L, Davis SM, Donnan GA, Parsons M. Tenecteplase versus Alteplase for Stroke Thrombolysis Evaluation Trial in the Ambulance (Mobile Stroke Unit-TASTE-A): protocol for a prospective randomised, open-label, blinded endpoint, phase II superiority trial of tenecteplase versus alteplase for ischaemic stroke patients presenting within 4.5 hours of symptom onset to the mobile stroke unit. BMJ Open. 2022 Apr 29;12(4):e056573. doi: 10.1136/bmjopen-2021-056573. PMID 35487712